CLINICAL TRIAL: NCT04198168
Title: The Predictive Performance of Renal Ultrasonographic Perfusion Measures on Changes in Renal Clearance in Response to Fluid Therapy.
Brief Title: The Predictive Performance of Renal Ultrasound on Changes in Renal Clearance
Status: Terminated | Type: Observational
Why Stopped: Due to the COVID-19 situation, it was not feasible to complete the study in our ICU.
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Johan Fridolf Hermansen, Principal Investigator, Aarhus University Hospital
Other Study IDs: 1-10-72-75-19
Record Dates: First submitted 2019-11-08; First posted 2019-12-13 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Acute Kidney Injury; Hypoperfusion; Fluid Overload
Keywords: Ultrasound; Renal perfusion; Fluid treatment; Venous congestion; Renal function
MeSH Terms: conditions — Acute Kidney Injury; Edema; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients: ICU patients who are assessed by their attending physician as having need for fluid therapy and are planned to receive IV crystalloid fluid due to oliguria and/or to improve GFR.
  Interventions: Drug: IV crystalloid fluid bolus

INTERVENTIONS:
Drug: IV crystalloid fluid bolus — The participant receives IV fluid as a standardised bolus of 7 ml/kg (ideal body weight).

SUMMARY:
The study will examine the ability of renal ultrasound (Doppler and Contrast Enhanced Ultrasound (CEUS)) in distinguishing ICU patients who exhibit increases in glomerular filtration rate (GFR) in response to fluid loading, from those for whom fluid loading is without benefit of directly harmful.

DETAILED DESCRIPTION:
The study will examine the ability of renal ultrasound (Doppler and Contrast Enhanced Ultrasound (CEUS)) in distinguishing ICU patients who exhibit increases in GFR in response to fluid loading, from those for whom fluid loading is without benefit of directly harmful.

Patients available for inclusion will receive a baseline administration of Tc-99-DTPA for precise determination of GFR/renal function by blood and urine samples.

Baseline values of ultrasound measures will be obtained, including renal arterial, renal venous, portal venous and hepatic venous Doppler measures and renal contrast enhanced ultrasound (CEUS) will also be recorded.

After two hours, baseline values of GFR are finished. The patient is then exposed to passive leg raising and ultrasound measures are repeated, including renal arterial, renal venous, portal venous and hepatic venous Doppler measures.

The participant then receives a standardised fluid bolus of 7 ml/kg (ideal body weight) Once the fluid bolus administration is complete, renal ultrasound is repeated, including renal arterial, renal venous, portal venous, hepatic venous Doppler measures and renal CEUS.

Follow-up determination of GFR/renal function based on Tc-99-DTPA after fluid therapy is repeated with blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years admitted to the ICU, Aarhus University Hospital.
* Patients who are assessed by their attending physician as having need for fluid therapy.

Exclusion Criteria:

* Insufficient ultrasound imaging of the kidneys.
* Pregnancy.
* Intolerance to any ultrasound contrast agent or isotopes, including intolerance for human albumin.
* Prior enrolment in a conflicting research study.
* Known morphological kidney disease.
* Need for dialysis.
* Need for extracorporeal membrane oxygenation (ECMO).
* Prior participation.
* Severe pulmonary hypertension (systolic pulmonary pressure > 90 mmHg)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU at Aarhus University Hospital
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in renal function in response to a standardised fluid bolus. | 6 hours
  Renal function is measures as Tc-99-Diethylenetriaminepentaacetic acid (DTPA) clearance.

SECONDARY OUTCOMES:
Renal venous flow classification | 6 hours
  normal - abnormal (pulsatile/biphasic/monophasic
Renal venous impedance index | 6 hours
  (maximum flow velocity - minimum diastolic flow velocity) / maximum flow velocity
Renal venous stasis index | 6 hours
  (index cardiac cycle time - venous flow time) / index cardiac cycle time
Renal arterial resistive index | 6 hours
  (maximum flow velocity - minimum diastolic flow velocity) / maximum flow velocity
Portal venous pulsatility fraction | 6 hours
  (maximum flow velocity - minimum diastolic flow velocity) / maximum flow velocity
Contrast enhanced ultrasound 1 | 6 hours
  Mean transit time (mTT)
Contrast enhanced ultrasound 2 | 6 hours
  Perfusion Index (PI)
Contrast enhanced ultrasound 3 | 6 hours
  Relative Blood Volume (rBV)
Contrast enhanced ultrasound 4 | 6 hours
  Wash-in Rate (WiR)
Contrast enhanced ultrasound 5 | 6 hours
  Quality Of Fit (QOF)
Continuous recordings of hemodynamic variables 1 | 6 hours
  arterial pressure
Continuous recordings of hemodynamic variables 2 | 6 hours
  Central venous pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Department of Anaesthesiology, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No